CLINICAL TRIAL: NCT01256203
Title: Prospective, Randomized, Controlled, Partially Blinded, Skin Photobiological Clinical Study of the Efficacy and Safety of a Sunscreen Product as Skin Protector Against Porfimer Sodium-induced Phototoxicity to Visible Light
Brief Title: Efficacy and Safety of a Sunscreen Against Porfimer Sodium-induced Phototoxicity to Visible Light
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor cancelled the study
Sponsor: Pinnacle Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: MA-PO-PHOTB05-01
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: High-grade Dysplasia in Barrett Esophagus; Non Small Cell Lung Cancer; Esophageal Cancer
Keywords: PDT; Porfimer sodium; Phototoxicity; Sunscreen
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Dermatitis, Phototoxic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunscreen (Experimental): Solar Protection Formula SPF® 60 will be applied on the skin of each subject. Applications will be followed by photobiological testings to assess skin protection.
  Interventions: Drug: Solar Protection Formula SPF® 60; Procedure: Photobiological testing

INTERVENTIONS:
Drug: Solar Protection Formula SPF® 60 — Solar Protection Formula SPF® 60 (2 mg/cm²) will be topically applied on a randomly predetermined specific skin area on the back of each subject on four separate occasions over 3 months. The same skin area will never be exposed more than once to the sunscreen.
Procedure: Photobiological testing — Photobiological testing will consist of exposing a small area of the sunscreen-protected and unprotected (control) skin areas to visible light on four separate occasions over 3 months. Light will be applied 30 minutes after application of the sunscreen. The same skin area will never be exposed more than once to light.

SUMMARY:
Photodynamic therapy (PDT) uses a combination of a drug, porfimer sodium, and a light from a non heated laser. The activation of the drug is done by illuminating abnormal areas using a fiber optic device. The fiber optic device is a very fine fiber (like fishing line) that permits transmission of light. By itself, porfimer sodium is inactive. However it becomes active when it is put in the presence of a light source such as sunlight, very intense indoor light, or laser. Therefore, the main risk with this therapy is that the skin will be more sensitive to light, and this sensibility can last up to 90 days. The skin reaction is similar to sunburn and is called phototoxicity.

To date, no product on the market has shown protection against visible light, and therefore, no product has been demonstrated to protect against the skin phototoxicity to visible light. A sunscreen sold under the brand name Solar Protection Formula® SPF 60 in the United States contains ingredients that provide maximum ultraviolet (UV) protection, as well as a formulation that could provide visible light protection. The product could potentially prevent the skin phototoxicity due to visible light, the most frequently reported side effect in patients receiving PDT with porfimer sodium. Therefore, this study is designed to assess the efficacy of topical application of Solar Protection Formula® SPF 60 as skin protector against visible light-induced skin redness and swelling following injection of porfimer sodium. It will involve 17 to 20 human subjects in the United States for whom PDT with porfimer sodium is planned for the treatment of high-grade dysplasia in Barrett's esophagus (pre-cancerous change in the food pipe tissue), lung cancer, or cancer of the esophagus (food pipe).

DETAILED DESCRIPTION:
Human subjects with planned PDT course will be evaluated to confirm eligibility. Prior to enrollment, all inclusion and exclusion criteria will be verified. Medical procedures including demographic information (age, sex, race, smoking and drinking habits), medical/surgical history, physical exam (including vital signs, body weight, height, and skin color), clinical laboratory testing, concomitant medication intake and other therapy uses will be collected. The study procedures will begin after the intravenous injection of porfimer sodium.

Skin photobiological testing will consist of four 2-day periods performed over three months after the injection of porfimer sodium at a dose of 2 mg/kg of body weight. Each period will include a Skin Illumination session and a Skin Evaluation session. During the Skin Illumination session, the Solar Protection Formula® SPF 60 will be randomly applied at a dose of 2 mg/cm² on a skin subunit area of the back 30 minutes before illumination. A second skin subunit will be used as a "no-treatment" observational area. Therefore, each subject will be her/his own control. Illumination will be performed using a visible light source. During the Skin Evaluation session, skin reactions will be scored by an outcome assessor 24 hours after illumination according to a pre-determined rating scale. The outcome assessor will be blinded to the active treatment sequence applications. All subjects will be followed for three months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are males or females aged 18 or older.
* Subjects scheduled to undergo PDT with porfimer sodium for an approved indication.
* Fair-skin human subjects with skin types II or III (blond or red hair, freckles, blue or green eyes) according to Fitzpatrick Classification.
* Subjects must be entirely free of any vitamin A, provitamin A, beta-carotene supplements, or photosensitizing agents, taken orally or topically applied on the back area to be used for the skin photobiological testing procedures, for at least 30 days prior to the injection of porfimer sodium.
* Non-menopausal or non-sterile female subjects of childbearing potential must have a negative pregnancy test at the time of entry into the study.
* Non-menopausal or non-surgically sterilized female subjects of childbearing potential must use a medically acceptable form of birth control.
* Subjects must sign an Informed Consent Form, which must comply with the International Conference on Harmonisation (ICH) guidelines and local requirements.

Exclusion Criteria:

* Subjects who have received PDT during the six months prior to the date of the informed consent signature.
* Subjects who would likely need a second PDT course within 90 days.
* Subjects with clinically significant skin disorders, particularly in the back areas to be used for the skin photobiological testing procedures.
* Subjects with intensive pigmented skin, pre-existing redness, or significant growth of hair in the back area to be used for the skin photobiological testing procedures.
* Subjects with a presence or history of skin neoplasms.
* Subjects with jaundice or porphyria cutanea tarda.
* Subjects with frequent manifestations of vasomotor instability with flushing.
* Subjects suffering from end-stage malignancy.
* Known porphyria or hypersensitivity to sunlight or intense artificial light.
* Known contraindications or hypersensitivity/allergy to excipients contained in the sunscreen formula.
* Subjects with severe acute respiratory distress caused by an obstructing endobronchial lesion.
* Subjects with a presence or history of neoplasms (treated during the last five years prior to study entry) other than carcinoma in situ of the cervix.
* Subjects with esophageal or gastric varices.
* Subjects with severe renal or hepatic impairment.
* Subjects with tracheoesophageal or bronchoesophageal fistula.
* Subjects with tumors eroding into a major blood vessel.
* Known contraindications or hypersensitivity/allergy to porfimer sodium.
* Subjects with esophageal ulcers > 1 cm in diameter.
* Female subjects who intend to become pregnant or intend to breast-feed during this study.
* Subjects unable to attend all visits required for the skin photobiological testing procedures.
* Subjects who have been treated with any investigational drug during 60 days prior to the date of the informed consent signature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Skin erythema responses of control (unprotected) and Solar Protection Formula® SPF 60-protected sites to light exposure | 17 days
  Skin erythema responses will be scored 24 hours after photobiological testing

SECONDARY OUTCOMES:
Skin erythema responses of control (unprotected) and Solar Protection Formula® SPF 60-protected sites to light exposure | 3 months
  Skin erythema responses will be scored 24 hours after photobiological testing on three separate occasions over 3 months
Skin edema responses of control (unprotected) and Solar Protection Formula® SPF 60-protected sites to light exposure | 3 months
  Skin edema responses will be scored 24 hours after photobiological testing on four separate occasions over 3 months
Skin phototoxicity responses of control (unprotected) and Solar Protection Formula® SPF 60-protected sites to light exposure | 3 months
  Skin phototoxicity responses will be scored according to the Common Terminology Criteria for Adverse Events (CTCAE) 24 hours after photobiological testing on four separate occasions over 3 months
Proportion of subjects with adverse events as a measure of safety | 3 months